CLINICAL TRIAL: NCT04847713
Title: Early Detection and Follow-Up of Patients With Fabry's Disease: New Biomarkers Approach
Brief Title: Early Detection and Follow-Up of Patients With Fabry's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Alvaro Hermida (Co-IP) (Unknown); Susana Belen Bravo (Unknown); Maria Teresa Cardoso (Unknown); Cristobal Colon Mejeras (Unknown); Maria Jose de Castro (Unknown); Emiliano Gonzalez-Vioque (Unknown); Elisa Leal Teles (Unknown); Saida Ortolano (Unknown); Jose Victor Alvarez (Unknown)
Responsible Party: Principal Investigator, Maria Luz Couce Pico, Head of neonatal department, Hospital Clinico Universitario de Santiago
Other Study IDs: CouFabry
Record Dates: First submitted 2021-03-26; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Fabry's Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fabry's disease: children and adults male or female between 6 and 70 years old, patients with diagnosis of FD, treated and non-treated
  Interventions: Other: extraction of blood samples
- Healthy controls: age and sex-matched group of healthy subjects with a negative family history for lysosomal storage disorders and no clinical signs of FD.
  Interventions: Other: extraction of blood samples

INTERVENTIONS:
Other: extraction of blood samples — Two blood samples (3.5 ml each) will be collected directly into purple K2-EDTA tubes and stored at 4°C for up to 24 hours for analysis

SUMMARY:
This research project will serve on the enhancement of early detection, diagnosis and follow-up of patients with Fabry Disease, through new biomarkers identification. This could have straight clinical impact on:

1. Early diagnosis, follow-up, and prediction of treatment response.
2. Suggestion about the optimal time to start treatment.
3. The data obtained will help to deepen our knowledge of the correlation among Lyso-Gb3, genotype and phenotype.
4. Better understanding of the pathophysiology of FD. To sum up, the results of the study will make a significant contribution to scientific knowledge providing new evidence with an immediate clinical application in FD patients.

As well as, the project will serve as the basis for a large-scale project implementation to validate the results obtained

DETAILED DESCRIPTION:
The overall purpose of the study is to identify biomarkers for FD in order to improve early detection and diagnosis, define pathological phenotypes and facilitate the monitoring of the disease and its response to therapy.

4.1 Primary objective o Identification of biomarkers for FD, mainly linked with phenotype (classic vs late onset); clinical manifestations (renal, cardiac and cerebrovascular FD associated complications) and treatment response.

4.2 Secondary objective o Correlate proteomic and transcriptomic data with geno-phenotype and especially with Lyso-Gb3 levels.

5 Methods

5.1 Study design This clinical study is an international, multicenter, prospective, open, with control group protocol, collecting biological samples (blood plasma) in patients diagnosed with FD (treated and non-treated patients) and healthy subjects. The same procedures will be done both control and FD patients.

All participants will be recruited during 15 months and all procedures will be placed over a single visit. The study will include two groups:

* FD patients (treated and untreated)
* Healthy controls

This study will be carried out with 3'omics analytical platforms (metabolomics, transcriptomics and proteomics) will be applied. Patients will be recruited through the Association of Lysosomal Patients-MPS Spain and Portugal and clinicians from Expert Centers in Spain and Portugal in this disorder. Children and adults of both sexes with a diagnosis of FD are eligible (refer to Section 5.2.1 Inclusion criteria).

This study will be performed in accordance with guidelines approved by the Galician (Spain) and Portuguese Ethics Committees. Expressed consent from patients or legal guardian/legal representative members if available will be written indicating that they understand the purpose and the procedures required for the study and are willing to participate in the study.

The informed consent must be obtained before performance of any study-related activity.

Information related to the following variables will be collected from each subject: age, sex, age at diagnosis, clinical symptoms at diagnosis, time of evolution, concomitant medications and start date, genetic study, lyso-Gb3 levels and α-GalA enzymatic activity. Blood samples (EDTA anti-coagulated, PAXgene Blood RNA, and Serum tubes) from each centre will be sent to our laboratory for proteomic and transcriptomic research assessment. If subjects are under ERT for FD, preinfusion and postinfusion samples will be obtained.

Disease diagnosis and phenotype will be classified as classic or later onset according internationally established criteria [17,18]. Recruited patients can be included in the study without receiving prior treatment or with some of the pharmacological alternatives authorized for commercialization, either replacement enzyme therapy and/or pharmacological chaperones. The same evaluations will also be carried out in healthy agesex matched controls.

5.2 Study Population

The study will obtain biological samples (one sample of blood plasma per participant) from patients with diagnosis of FD, treated and non-treated, recruited through the Association of Lysosomal Patients-MPS Spain and Portugal and clinicians from Expert Centres in Spain and Portugal in this disorder. An age and sex-matched group of healthy subjects will serve as controls. Controls will be identified from volunteers and nonmedical staff at the Clinical Hospital University of Santiago. Controls will be required to have a negative family history for lysosomal storage disorders and no clinical signs of FD.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: children and adults male or female between 6 and 70 years old.
2. Patients or legal representative will be able to give written informed consent. Parent(s) or guardian(s), for subject under 18 years of age, must be willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure.
3. Patients with diagnosis biochemically confirmed by a decrease in the enzymatic activity of alpha-galactosidase or genetically by the presence of a pathogenic variant in GLA
4. Controls: male or female subjects between 6 and 70 years old must be unaffected with Fabry Disease, and considered healthy with no previous history of diabetes mellitus, atherosclerotic vasculopathy or other inflammatory disease.

Exclusion Criteria:

1. Subject with inconclusive genetic diagnosis (i.e. carriers of variants of unknown significance (VUS) or variants with conflicting interpretations of pathogenicity).
2. Subject with any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to give his/her informed consent.
3. Subject or legal representative unable to or unwilling to give informed consent.
4. Subject participating in a study with an investigational drug within 3 months before consent.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Population The study will obtain biological samples (one sample of blood plasma per participant) from patients with diagnosis of FD, treated and non-treated, recruited through the Association of Lysosomal Patients-MPS Spain and Portugal and clinicians from Expert Centres in Spain and Portugal in this disorder. An age and sex-matched group of healthy subjects will serve as controls. Controls will be identified from volunteers and nonmedical staff at the Clinical Hospital University of Santiago. Controls will be required to have a negative family history for lysosomal storage disorders and no clinical signs of FD.
  The same procedures will be done both control and FD patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative proteomic analysis | 3 months
  will identifiy all the proteins expressed in all samples. Functional and quantitative analysis in each group will be performed by FunRich software, String, Reactome and a label free approach (SWATH-MS; Sequential Window Acquisition of all Theoretical Mass Spectra). Information about the change of each protein will be made by MARKERVIEW software
Transcriptomic study | 3 months
  includes sequencing of RNA libraries. FASTQ files will be analyzed by quantification of transcript expression using Salmon algorithm; correlation analysis and number of reads in each group with DESeq2 program obtaining PCA plot, p-value histogram, MA plot, Volcano Plot and correlation heatmap.
Integrative analysis of Omics | 6 months
  will only considere transcripts relatively high-correlated or anti-correlated with proteins of interest in the data. Global Spearman's correlations will be calculated between proteomic and transcript in each group

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luz Couce-Pico, MD, Principal Investigator — University Hospital of Santiago de Compostela
Locations (1):
- University Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No